CLINICAL TRIAL: NCT04909281
Title: Feasibility of Sending a Direct Send HPV Self-sampling Kit to Long-term Non-attenders in an Organized Cervical Screening Program
Brief Title: Feasibility of Sending a Direct Send HPV Self-sampling Kit to Long-term Screening Non-attenders
Status: Completed | Type: Observational
Sponsor: Falu Hospital (Other)
Responsible Party: Principal Investigator, Hanna Sahlgren, Principal Investigator, Falu Hospital
Other Study IDs: DNR 2019-02564
Record Dates: First submitted 2021-05-27; First posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: HPV; Cervical Cancer
Keywords: self sampling
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Long-term non-attenders in the cervical screening program: All women who had not attended tthe cervical screening program in Sweden for at least 10 years were eligeble.
  Interventions: Diagnostic Test: Self-sampling HPV

INTERVENTIONS:
Diagnostic Test: Self-sampling HPV — In this cohort study nested in the organized cervical screening program, all women who had not participated in the organized screening program for at least 10 years in one Swedish county were eligible.

SUMMARY:
All women in one Swedish county who had not participated in the organized screening program for at least 10 years were sent an HPV self-sampling kit. Women who were positive for HPV were referred to a gynecological examination including colposcopy and further testing according to national guidelines.

DETAILED DESCRIPTION:
In this cohort study nested in the organized cervical screening program, all women who had not participated in the organized screening program for at least 10 years in one Swedish county were eligible. Women were identified through the screening hub register that administrates for all invitations, referrals, and monitoring of the cervical screening program. The county screening hub invites approximately 30 000 women yearly to routine screening. Those who had opted out of the screening program, undergone hysterectomy, or changed their personal identification number (PNR) were excluded. HPV self-sampling kits with instructions and invitation letters were sent from the Department of Laboratory Medicine, Falun Hospital, in batches over 4 weeks. Lists of invitees were checked against changes in the screening hub register for individuals who moved, emigrated, died, or had taken a routine screening sample before sending a kit. Samples were received and HPV-analysis was performed.

If the self-sample HPV test was negative, the woman was returned to the screening program according to routine practice. HPV-positive women were referred without triage for further investigation to a gynecologist responsible for the clinical follow-up of high-risk women. The gynecological examination included colposcopy as well as biopsies and a liquid based cytology (LBC) sample (analyzed for cytology and HPV), which are routine examinations in clinical practice according to national and international guidelines. Colposcopies were performed within 3 months of a positive self-sample. If the colposcopic examination or the cytological/histopathological results indicated high-grade squamous intraepithelial lesions (HSIL) or invasive cervical cancer, women underwent treatment by conization and/or hysterectomy according to national guidelines The Cobas® PCR Female Swab Sample Packet was used for self-sampling, as previous studies had determined that the sensitivity for HPV was high and comparable with cervical samples used in the organized screening program. The HPV analysis was performed at the Department of Laboratory Medicine, Falun Hospital using the Cobas 4800 HPV Test (Roche Molecular Systems, South Branchburg, New Jersey, USA).

ELIGIBILITY:
Inclusion Criteria:

- Women who had not participated in the organized screening program for at least 10 years

Exclusion Criteria:

- Women who were hystrectomized, moved, died

Ages: 33 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women get cervical cancer
Study Population: Women who had not participated in the organized screening program for at least 10 years in 1 Swedish county
Sampling Method: Probability Sample
Enrollment: 741 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2020-04-04 (Actual)

PRIMARY OUTCOMES:
Histopathologically confirmed high grade cervical lesions and cervical cancer among long-trem non-attenders in the organized cervical screening program | 1 year
  To evaluate the prevalence of high grade cervical lesions and cervical cancer cancer among long-term non-attenders in the organized screening program

CONTACTS AND LOCATIONS:
Overall Officials: Hanna I Sahlgren, md, Principal Investigator — RCC; Miriam K Elfström, phd, Principal Investigator — RCC
Locations (1):
- Falu Lasarett, Falun, Dalarna County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Share upon demand
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 years
Access Criteria: Contact principal investigator